CLINICAL TRIAL: NCT01251835
Title: A Phase 1, Open Label, Fixed Sequence Design, Multiple Dose Study To Assess The Effect Of Rifampin On The Pharmacokinetics Of Sitaxsentan In Healthy Subjects
Brief Title: Effect Of Rifampin On Pharmacokinetics Of Sitaxsentan
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1321060
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2011-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Sitaxsentan; Rifampin; Drug Interaction; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — sitaxsentan; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitaxsentan (Active Comparator)
  Interventions: Drug: Sitaxsentan alone
- Sitaxsentan plus Rifampin (Experimental)
  Interventions: Drug: Sitaxsentan; Drug: Rifampin

INTERVENTIONS:
Drug: Sitaxsentan alone — Days 1-5: Sitaxsentan tablet, 100 mg, q24 h (once a day)
  Arms: Sitaxsentan
Drug: Sitaxsentan — Days 6-12: Sitaxsentan tablet, 100 mg, q24h (once a day)
  Arms: Sitaxsentan plus Rifampin
Drug: Rifampin — Days 6-12: Rifampin capsule, 600 mg, q24h (once a day)
  Arms: Sitaxsentan plus Rifampin

SUMMARY:
This study will assess how rifampin will affect the blood levels of sitaxsentan. Safety of sitaxsentan given alone and with rifampin will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or women of non-child bearing potential.
* Subjects between the ages of 21 and 55 years, inclusive.
* Signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Has hepatic dysfunction.
* Has history of excessive alcohol and tobacco use.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Peak Plasma Concentrations of sitaxsentan co-administered with rifampin versus sitaxsentan administered alone. | 24 hours
Comparison of Area Under the Curve of sitaxsentan co-administered with rifampin versus sitaxsentan administered alone. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321060&StudyName=Effect%20Of%20Rifampin%20On%20Pharmacokinetics%20Of%20Sitaxsentan